CLINICAL TRIAL: NCT06124430
Title: Effect of Using the ECOX Teaching Tool in the Emergency Department on OSCEs for Medical Students: Randomized Controlled Trial
Brief Title: Emergency Structured Clinical Examination Training bOX
Acronym: ECOX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, DENISE JOLIVOT, Responsable DRCI, University Hospital, Angers
Other Study IDs: 202300116
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Students will take part in the ECOS of the departments scheduled at the end of their internship. Students will use the various revision methods usually offered to them by the faculty or in the emergency department, apart from the ECOX tool. Revision methods are left to their own discretion.
- ECOX Interventional Group: Students will take part in the ECOS of the departments scheduled at the end of their internship. Students will use the ECOX tool available in the emergency department to practice before taking the on-duty OSCEs.
  Interventions: Other: ECOX box

INTERVENTIONS:
Other: ECOX box — For the ECOX approach, they will have the various ECOX grids and a stopwatch at their disposal in the 2 units of the emergency department. There will be around thirty evaluation grids at their disposal. Students will choose the ECOX grid corresponding to a starting situation. Once the time limit has elapsed, they must compare their answers with the grid's expectations. Each completed grid will be returned to a drawer in the box, to assess adherence to the tool and suggestions for grid modifications, as well as any comments. Students will be able to use them as many times as they wish during the course and before the service ECOS.
  Groups: ECOX Interventional Group

SUMMARY:
This is a pragmatic, randomized, controlled study carried out in the emergency department of Angers University Hospital.

All students on placement over a 10-week period will be able to take part in the study. After a clear explanation to the students during the welcome meeting, followed by the collection of free and informed non-opposition, the students will be assigned according to the "ECOX" or "traditional" approach, depending on the randomization status of the internship period. The inclusion arm will be the same for all students over the placement period.

For the traditional approach (control group), students will participate in the OSCEs of the services scheduled at the end of the internship. Students will use the various revision methods usually offered to them by the faculty or in the emergency department, apart from the "ECOX tool". Revision methods are left to their own discretion. Students will complete the internship without any knowledge of the ECOX tool.

For the ECOX approach, students included in the intervention arm will be invited to use the ECOX tool. They will have the various ECOX grids and a stopwatch at their disposal in the 2 units of the emergency department. They will have around thirty evaluation grids at their disposal. The students will choose the ECOX grid corresponding to their initial situation, based on the nurse's triage of the patient. They must ask the patient's permission to practice with them. They must not look at the ECOX grid. As with the on-duty ECOS, they will have 7 minutes to complete the interview and clinical examination. Once this time has elapsed, they will have to compare their answers with the expectations of the grid. They may also be observed by a co-external study participant, a department intern or a senior staff member who is not involved in the OSCE evaluation. They will act as observers and complete the grid. The students will then be able to propose modifications to the grids. Each completed grid will be returned to a drawer in the cubicle, to assess adherence to the tool and suggestions for grid modifications, as well as any comments.

Students will be able to use them as many times as they like during the course and before the service ECOS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Medical student in a non-ERASMUS emergency department
* Participating in the service ECOS planned at the end of the internship
* No free and informed consent from the student.

Exclusion Criteria:

* Refusal to participate in the study.
* Student returning to the emergency department and having already participated in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students present during their internship in the emergency department will be offered the opportunity to take part in a study of educational research in the emergency department.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-11-07 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the value of the ECOX tool in improving the final grade for service ECOS compared with standard learning during the training course. | 10 weeks
  the students' average score on the end-of-course OSCEs. This criterion will correspond to the average of all students per arm, who passed the same OSCE stations from one course to the next.

SECONDARY OUTCOMES:
Describing the ECOX tool versus control of psychological status prior to ECOS | 10 weeks
  Average STAI-Y (State-Trait Anxiety) scores between the two groups.
Evaluate the ECOX tool versus control of student know-how | 10 weeks
  The average scores on the behavioral assessment during the service ECOS between the two groups.

IPD SHARING:
Plan to Share IPD: Undecided